CLINICAL TRIAL: NCT02378181
Title: Testing the Effectiveness of a Graphic Novel Health Education Curriculum for Patients With Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Treatment Research Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Organization: Public Health Management Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1411; CDR-1310-07308 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Results first posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2022-10

CONDITIONS: Alcohol Use; Drug Use
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Toolkit (TK) (Experimental): Patients in the TK condition will receive counseling sessions from participating counselors who have been trained to use the Health Education Toolkit (TK).
  Interventions: Behavioral: Health Education Toolkit
- Treatment-as-usual (TAU) (Active Comparator): Patients in the treatment-as-usual (TAU) condition will receive the same number of counseling sessions as patients in the TK condition from participating counselors who have not been trained to use the Health Education Toolkit. Counselors working with patients in this condition will receive a control training of the same length and intensity on recovery topics that are covered in the Health Education Toolkit, but will not be equipped with the Toolkit.
  Interventions: Behavioral: Treatment-as-usual

INTERVENTIONS:
Behavioral: Health Education Toolkit — An existing evidence-based toolkit intervention will be adapted and redesigned by a patient and provider team into an engaging, narrative graphic novel curriculum. The proven behavioral interventions will be augmented with health education material focused on MAT and HIV risk reduction. Together, these materials will comprise the Health Education Toolkit. The Health Education Toolkit (TK) will employ a shared decision making model to encourage 1) increased recovery engagement by patients, and 2) patient engagement in deciding whether to initiate and adhere to MAT.
  Arms: Toolkit (TK)
Behavioral: Treatment-as-usual — Treatment-as-usual will consist of the same number of counseling sessions as the experimental TK condition, but the counselors working with patients in this condition will not be equipped with the TK materials.
  Arms: Treatment-as-usual (TAU)

SUMMARY:
This study deploys a strategy to develop and evaluate a training-efficient, multimedia patient-centered Health Education Toolkit to promote shared decision making between counselors and patients. An existing evidence-based toolkit intervention will be adapted and redesigned by a patient and provider team into an engaging, narrative graphic novel curriculum useful in group and individual counseling. The proven behavioral interventions will be augmented with health education material focused on medication assisted treatment (MAT). We will assess feasibility and acceptability, and pilot test whether exposure to the Toolkit (TK) can shared decision making conversations, reduce substance use, and increase engagement with MAT.

DETAILED DESCRIPTION:
An existing evidence-based toolkit intervention will be adapted and redesigned by a patient and provider team into an engaging, narrative graphic novel curriculum useful in group and individual counseling. The proven behavioral interventions will be augmented with health education material focused on medication assisted treatment (MAT) and HIV risk reduction. Together, these materials will comprise the Health Education Toolkit. The Health Education Toolkit (TK) will employ a shared decision making model to encourage 1) increased recovery engagement by patients, and 2) patient engagement in deciding whether to initiate and adhere to MAT. We will conduct a randomized pilot trial of 50 patients with active alcohol substance use disorders (SUDs) enrolled in inpatient or outpatient treatment and will follow them over 3 months. We will test whether patients randomized to receive the TK curriculum will report increased shared decision making conversations, report greater satisfaction and acceptability of their treatment sessions, demonstrate larger reductions in substance use (drug and alcohol) and increases in abstinence, demonstrate improved alcohol severity scores, attend more attendance at specialty substance abuse intervention and treatment sessions, and demonstrate greater rates of initiating MAT for alcohol dependence over the 3-month follow-up period as compared to patients receiving treatment-as-usual (TAU).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Screening score of at least 16 on the AUDIT
* Meets criteria for a DSM-V substance use disorder as assessed via the MINI Plus 5.0.
* Reports at least two heavy drinking episodes in the previous 4 weeks

Exclusion Criteria:

* Reports plans to leave the Philadelphia greater metropolitan area within the next 6 months
* Does not speak English
* Unable to provide valid informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam C Brooks, PhD, Principal Investigator — Treatment Research Institute
Locations (2):
- United States (2):
  - Wedge Medical Center, Philadelphia, Pennsylvania
  - Kirkbride Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Patient-Centered Outcomes Research Institute (PCORI) Project Abstract — http://www.pcori.org/research-results/2014/testing-effectiveness-graphic-novel-health-education-curriculum-patients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from addiction treatment programs in the Philadelphia region between August 2016 and January 2017
Pre-assignment Details: Participants were screened for eligibility using the AUDIT and Mini-International Neuropsychiatric Interview (MINI) for substance use disorders.
Period: Overall Study
Arm/Group | Toolkit (TK) | Treatment-as-usual (TAU)
Started | 21 | 28
6 Week Assessment | 18 | 16
3 Month Assessment | 18 | 21
Completed | 18 | 21
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Incarcerated | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who completed the baseline assessment and randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Toolkit (TK) | Treatment-as-usual (TAU) | Total
Number analyzed (Participants) | 21 | 28 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 28 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.71 (10.26) | 43.30 (10.63) | 43.04 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number analyzed differs from overall because one participant's sex is unknown
  Participants
    number analyzed (Participants) | 21 | 27 | 48
    Female | 6 | 11 | 17
    Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 18 | 24 | 42
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 14 | 30
  White | 3 | 9 | 12
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: Participants]
  United States | 21 | 28 | 49

OUTCOME MEASURES:

1. Primary Outcome: Shared Decision Making Conversations, as Measured by the Shared Decision Making Questionnaire (SDM-Q)
Description: Shared decision making score, as measured by the Shared Decision Making Questionnaire (SDM-Q) which uses a 1-6 point scale with higher numbers indicating greater shared decision-making. Results are presented for one research site only because of counselor randomization issues at the second site (i.e., the randomization was extremely unbalanced with 7 TAU counselors and 1 TK counselor).
Time Frame: 3 months
Population: Patients who completed the 3-month follow-up at one research site.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Toolkit (TK) | Treatment-as-usual (TAU)
Number analyzed (Participants) | 17 | 12
units on a scale | 5.14 (0.78) | 4.55 (1.34)

2. Primary Outcome: Treatment Satisfaction and Acceptability, as Measured by the Satisfaction Survey
Description: Satisfaction and acceptability of treatment sessions measured on a 1-5 scale with higher scores indicating greater satisfaction. Results are presented for one research site only because of counselor randomization issues at the second site (i.e., the randomization was extremely unbalanced with 7 TAU counselors and 1 TK counselor).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Toolkit (TK) | Treatment-as-usual (TAU)
Number analyzed (Participants) | 17 | 13
units on a scale | 3.95 (.86) | 3.97 (1.14)

3. Secondary Outcome: Substance Use, as Measured by the Timeline Followback and Confirmed by Urinalysis
Description: Days substance use as measured by the Timeline Followback and confirmed by urinalysis. Results are presented for one research site only because of counselor randomization issues at the second site (i.e., the randomization was extremely unbalanced with 7 TAU counselors and 1 TK counselor).
Time Frame: 3 months
Population: Participants who completed the 3-month follow-up at one research site
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Toolkit (TK) | Treatment-as-usual (TAU)
Number analyzed (Participants) | 16 | 11
Days
  Used Alcohol | 12.00 (14.53) | 22.91 (27.08)
  Used Drugs: number analyzed (Participants) | 15 | 11
  Used Drugs | 3.40 (5.77) | 1.27 (1.90)

4. Secondary Outcome: Substance Abuse Treatment Session Attendance, as Measured by the Non-Study Medical and Other Services (NSMOS)
Description: Self-reported days attended treatment for alcohol or drug use issues as measured by the Non-Study Medical and Other Services (NSMOS). Results are presented for one research site only because of counselor randomization issues at the second site (i.e., the randomization was extremely unbalanced with 7 TAU counselors and 1 TK counselor).
Time Frame: 6 weeks, 3 months
Population: The number of participants analyzed for the 6 week follow-up differs from the overall number analyzed because some participants did not complete the 6 week follow-up, but did complete the 3 month follow-up.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Toolkit (TK) | Treatment-as-usual (TAU)
Number analyzed (Participants) | 17 | 13
Days
  6 week follow-up: number analyzed (Participants) | 16 | 10
  6 week follow-up | 17.69 (11.56) | 15.60 (8.42)
  3 month follow-up | 10.69 (8.75) | 12.83 (17.68)

5. Secondary Outcome: Medication Assisted Treatment (MAT) Initiation, as Measured by a Utilization Review
Description: Initiation of MAT as measured by a chart utilization review. Results are presented for one research site only because of counselor randomization issues at the second site (i.e., the randomization was extremely unbalanced with 7 TAU counselors and 1 TK counselor).
Time Frame: 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Toolkit (TK) | Treatment-as-usual (TAU)
Number analyzed (Participants) | 17 | 13
percentage of participants | 0 | 8.3

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from each participant over a 6-month period of time.
Description: The study serious adverse event (SAE) definition did not consider pre-planned elective procedures and unrelated medical events that require hospitalization SAEs. Adverse events (AEs) that were not clinically significant (e.g., colds, other medical conditions not related to drug use) were not considered AEs. This reporting strategy was approved by the Institution Review Board overseeing the study and the funding agency.
Arm/Group | Toolkit (TK) | Treatment-as-usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/28
Other Adverse Events (participants affected / at risk) | 0/21 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Toolkit (TK) (N=21) | Treatment-as-usual (TAU) (N=28)
Hospitalization for Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT02378181/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT02378181/SAP_001.pdf